CLINICAL TRIAL: NCT05643807
Title: Bladder Washing Cytology for Detection of Urothelial Carcinoma Using Catheter or Flexible Cystoscope: Which is Better? A Prospective Randomized Study
Brief Title: Bladder Washing Cytology for Detection of Urothelial Carcinoma Using Catheter or Flexible Cystoscope: Which is Better?
Acronym: BWash
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Ilaria Lucca, Principal investigator, MD, Centre Hospitalier Universitaire Vaudois
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021-01124
Record Dates: First submitted 2022-11-21; First posted 2022-12-09 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Bladder Cancer
Keywords: Bladder cancer; Urinary cytology
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Urinary Catheters

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- urinary catheter (Active Comparator): Urinary cytology will be collected using a Ch.14 bladder catheter after the removal of the cystoscope. Catheter will be placed at the bladder neck level.
  Interventions: Device: Urinary catheter
- flexible cystoscope (Active Comparator): Urinary cytology will be collected through the flexible cystoscope itself at the end the cystoscopy. Before starting the urinary collection, the cystoscope will either be placed in front of a suspected intravesical lesion (if present) or at the bladder neck (if no lesion present).
  Interventions: Device: Flexible cystoscopy

INTERVENTIONS:
Device: Flexible cystoscopy — Urinary cytology will be collected through the flexible cystoscope itself at the end the cystoscopy. Before starting the urinary collection, the cystoscope will either be placed in front of a suspected intravesical lesion (if present) or at the bladder neck (if no lesion present).
  Arms: flexible cystoscope
Device: Urinary catheter — Urinary cytology will be collected through a Ch14 urinary catheter after the cystoscopy
  Arms: urinary catheter

SUMMARY:
Urine cytology can be collected with spontaneous urine or by washing the bladder. It is commonly accepted among urologist that instrumental bladder washing is the method of choice. There are, however, no solid recommendations regarding the method to collect the urine for bladder wash cytology during cystoscopy. There are mainly two possibilities: 1) the use of an intermittent bladder catheter after the removal of the cystoscope or 2) bladder lavage through working channel of the flexible cystoscope itself. The first choice may increase the number of collected cells because of the larger caliber of the catheter compared to the working channel and thus the better efficacy of bladder wash. However, this method is certainly more invasive and possibly more expensive. To the best of our knowledge and according to available literature, none of both collection method can be defined as gold standard. The aim of the study is to show that use of flexible cystoscope brings the same results in terms of quality of the urine collection for analysis as the use of intermittent bladder catheter and is less unpleasant for the patient. If our study confirms the non-inferiority of "direct" collection through the cystoscope, this will allow the establishment of recommendations in this sense in order to simplify the procedure and reduce as much as possible the manipulations within the urogenital tract.

DETAILED DESCRIPTION:
The aim of the study is to show that use of flexible cystoscope brings the same results in terms of quality of the urine collection for analysis as the use of intermittent bladder catheter and is less unpleasant for the patient.

Group A: Urinary cytology will be collected using a Ch.14 bladder catheter after the removal of the cystoscope. Catheter will be placed at the bladder neck level.

Group B: Urinary cytology will be collected through the flexible cystoscope itself at the end the cystoscopy. Before starting the urinary collection, the cystoscope will either be placed in front of a suspected intravesical lesion (if present) or at the bladder neck (if no lesion present).

ELIGIBILITY:
Inclusion Criteria:

1. Men aged > or = 18 years
2. Patients scheduled for a flexible cystoscopy and urinary cytology.
3. Patients who have signed the informed consent.
4. Patients who speak French

Exclusion Criteria:

1. Manipulations or instrumentation of urinary tract, including but not limited to Double-J stent placement or removal, and/or bladder biopsy
2. Inability to give informed consent or without capacity of discernment

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Enrollment: 414 (Estimated)
Dates: Start 2023-02-08 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
The quality of urinary cytology according to the tool used for collection of both groups | 2 years
  Number of urothelial cells, number of inflammatory cells, presence of necrosis or blood will be used to assess this outcome measure

SECONDARY OUTCOMES:
The sensitivity and sensibility of the urinary cytology of both groups | 2 years
  Sensitivity ans specificity percentage will be calculated based on the results of both urinary cytology and cystoscopy
The satisfaction of patients of both groups | 2 years
  The Faces Pain Scale will be used for each patient after the cytology to assess his satisfaction/pain (0= no pain and 10=the worst pain possible)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire Vaudois, CHUV, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided